CLINICAL TRIAL: NCT00653549
Title: Comparative, Randomized, Single-Dose, 2 Way Cross Over Bioavailability Study of Par Torsemide Tablets 20mg With That of Roche Demadex 1*20 mg in Healthy Subjects Under Fasting Conditions.
Brief Title: Bioavailability Study of Torsemide Tablets Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Par Pharmaceutical, Inc. (Industry)
Collaborators: Anapharm (Industry)
Responsible Party: Dr. Alfred Elvin/ Director Biopharmaceutics, Par Pharmaceutical, Inc.
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 01169
Record Dates: First submitted 2008-04-01; First posted 2008-04-07 (Estimated); Last update posted 2011-06-17 (Estimated); Status verified 2011-06

CONDITIONS: To Determine Bioequivalence Under Fasting Conditions
Keywords: Bioequivalence; Torsemide Tablets; fasting
MeSH Terms: conditions — Fasting | interventions — Torsemide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Subjects received Par formulated product under fasting conditions
  Interventions: Drug: Torsemide
- B (Active Comparator): Subjects received Roche formulated product under fasting conditions
  Interventions: Drug: Demadex

INTERVENTIONS:
Drug: Torsemide — Tablets, 20 mg, single-dose
  Other Names: Demadex
  Arms: A
Drug: Demadex — tablets, 20 mg, single-dose
  Other Names: Torsemide
  Arms: B

SUMMARY:
To compare the single-dose bioavailability of Torsemide tablets with Demadex

DETAILED DESCRIPTION:
To compare the single -dose bioavailability of Par Torsemide tablets 20mg with that Roche Demadex 1*20mg tablets under fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

Subjects enrolled in the study will be members of the community at large.

* The Recruitment will be done by radio, newspapers and Anapharm Inc.
* Anapharm Website advertisements.
* Subjects must meet all the following criteria in order to be included in the study.
* Subjects will be male and / or female, smokers and non-smokers, 18 years of age and older.
* Subjects should read, sign, and date an Informed Consent form prior to the study procedures.
* Subjects must complete all screening procedures within 28 days prior to the administration of the study medication.

Exclusion Criteria:

* Breast- feeding female subjects.
* Any clinically significant abnormality found during medical screening.
* Subjects with BMI ≥30
* Any Clinically significant gastrointestinal pathology (e.g. chronic diarrhea, inflammatory bowel diseases) or unresolved gastrointestinal symptoms (e.g. diarrhea, vomiting), susceptible of interfering with the absorption of drugs.
* Clinically significant illness within 4 weeks prior to the administration of the study medication
* Abnormal laboratory tests judged clinically significant.
* ECG abnormalities (clinically significant) (PR interval greater than 225ms);or vital sign abnormalities (systolic blood pressure lower than 90 or over 140 mmHg, diastolic blood pressure lower than 60 or over 95 mmHg, or heart rate less than 60 bpm) at screening.
* History of allergic reactions to torsemide or sulfonylureas (e.g. tolbutamide, chlorpropamide, glyburide and gliclazide) or other related drugs ( e.g. furosemide, bumetanide, sulfabenzamide, sulfacetamide, sulfathiazole, sulfadiazine, sulfamethoxazole, sulfasalazine, sulfisoxazole and dapsone).
* Any food allergy, intolerance, restriction or special diet that, in the opinion of the Medical Sub- Investigator, could contraindicate the subject's participation in this study.
* Positive urine drug screen at screening.
* Positive testing for hepatitis B, hepatitis C, or HIV at screening.
* Positive urine pregnancy test at screening.(performed on all female subjects)
* Use of an investigational drug or participation in an investigational study within 30 days prior to administration of the study medication.
* Donation of plasma ( 500 mL) within 7 days or donation of significant loss of whole blood (450 mL) within 56 days prior to administration of the study medication.
* History of significant alcohol abuse within six months of the screening visit or any indication of the regular use of more than two units of alcohol per day (1 Unit = 150 mL of wine or 360 mL of beer or 45 ml of alcohol 40%)
* History of drug abuse or use of illegal drugs: Use of soft drugs (such as marijuana, pot) within 3 months of the screening visit or hard drugs (such as cocaine, phencyclidine [PCP] and crack) within 1 year of the screening visit.
* Subjects who have taken prescription medication within 14 days prior to administration of study medication or over the counter products within 7 days prior to administration of study medication, except for topical products without systemic absorption.
* Female subjects of childbearing potential having unprotected sexual intercourse with any non- sterile male partner (i.e. male who has not been sterilized by vasectomy for al least 6 months) within 14 days prior to study drug administration. The Acceptable methods of contraception are :
* Condom+ spermicide (within 14 days prior to study drug administration)
* Diaphragm + spermicide (within 14 days prior to study drug administration.
* Intrauterine contraceptive device (place al least 4 weeks prior to study drug administration)
* Subjects who have taken any drugs known to induce or inhibit hepatic drug metabolism within 30 days prior to administration of the study medication.
* (examples of inducers: barbiturates, carbamazepine, phenytoin,glucocorticoids, rifampin,rifabutin; examples of inhibitors: antidepressants, cimetidine, diltiazem, erythromycin, ketoconazole, MAO inhibitors, neuroleptics, verapamil, quinidine)
* Subjects who have undergone clinically significant surgery within 4 weeks prior to the administration of the study medication.
* Any reason which, in the opinion of the investigator, would Prevent the subject from participating in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2001-04; Primary Completion 2001-05 (Actual); Study Completion 2001-05 (Actual)

PRIMARY OUTCOMES:
Rate and Extend of Absorption | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Eric Masson, Principal Investigator — Anapharm